CLINICAL TRIAL: NCT03044158
Title: GeneXpert Performance Evaluation for Linkage to Tuberculosis Care: The XPEL-TB Trial
Brief Title: GeneXpert Performance Evaluation for Linkage to Tuberculosis Care
Acronym: XPEL-TB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Makerere University (Other); Johns Hopkins Bloomberg School of Public Health (Other); London School of Hygiene and Tropical Medicine (Other); Yale University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R01HL130192 (NIH); PACTR201610001763265 (Registry Identifier: Pan African Clinical Trials Registry); R01HL130192 (NIH)
Record Dates: First submitted 2017-01-23; First posted 2017-02-06 (Estimated); Results first posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-01

CONDITIONS: Tuberculosis, Pulmonary; Rifampicin Resistant Tuberculosis
Keywords: tuberculosis; implementation science; point-of-care; diagnostics; GeneXpert; Uganda
MeSH Terms: conditions — Tuberculosis, Pulmonary; Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Onsite ZN or LED fluorescence microscopy + hub-based GeneXpert testing per existing protocols
- Intervention (Experimental): Onsite molecular testing for TB with GeneXpert I + process redesign to facilitate same-day TB diagnosis and treatment + performance feedback
  Interventions: Device: GeneXpert I; Behavioral: Process re-design; Other: Performance Feedback

INTERVENTIONS:
Device: GeneXpert I — Onsite molecular testing with GeneXpert I as a replacement for microscopy
  Other Names: GeneXpert
  Arms: Intervention
Behavioral: Process re-design — Research and Uganda NTLP staff will engage health center staff in a discussion of how to re-organize clinical, laboratory and pharmacy services to enable same-day TB diagnosis and treatment.
  Arms: Intervention
Other: Performance Feedback — Feedback of TB diagnostic evaluation quality indicators to health center staff
  Arms: Intervention

SUMMARY:
The investigators' overall objective is to assess the effectiveness, implementation and costs of a streamlined TB diagnostic evaluation strategy based around rapid, onsite molecular testing. The intervention strategy was developed based on theory-informed assessment of barriers to TB diagnostic evaluation at community health centers in Uganda and a process of engagement with local stakeholders. It includes: 1) Point-of-care molecular testing using GeneXpert as a replacement for sputum smear microscopy; 2) Re-structuring of clinic-level procedures to facilitate same-day TB diagnosis and treatment; and 3) Quarterly feedback of TB evaluation metrics to health center staff. The investigators' central hypothesis is that the intervention strategy will have high uptake and increase the number of patients diagnosed with and treated for active pulmonary TB. To test this hypothesis, the investigators will conduct a pragmatic cluster-randomized trial at community health centers that provide TB microscopy services in Uganda in partnership with the National TB Program (NTP). The investigators utilize an effectiveness-implementation hybrid design in which, concurrent with the clinical trial, the investigators will conduct nested mixed methods, health economic and modeling studies to assess 1) whether the intervention strategy modifies targeted barriers to TB diagnostic evaluation; 2) fidelity of implementation of the intervention components (i.e, the degree to which intervention components were implemented as intended vs. adapted across sites); and 3) cost-effectiveness and public health impact.

DETAILED DESCRIPTION:
Aim 1: To compare patient outcomes at health centers randomized to intervention vs. standard-of-care TB diagnostic evaluation strategies. The investigators will randomize 20 community health centers to continue standard TB evaluation (routine microscopy plus referral of patients for Xpert testing per existing processes of care) or to implement the intervention strategy (1. Onsite molecular testing; 2. Re-structuring clinic-level procedures to facilitate same-day TB diagnosis and treatment; and 3. Performance feedback). The investigators will compare reach and effectiveness based on the numbers and proportions of patients (N=5500) who complete TB testing, are found to have TB, and have treatment initiated within one week of specimen provision.

Aim 2: To identify processes and contextual factors that influence the effectiveness and fidelity of the intervention TB diagnostic evaluation strategy. The investigators will use quantitative process metrics to assess the adoption and maintenance over time of the core components of the intervention strategy. The investigators will also collect quantitative and qualitative data to describe the fidelity of implementation of each component and faithfulness to the conceptual model.

Aim 3: To compare the costs and epidemiological impact of intervention vs. standard-of-care TB diagnostic evaluation strategies. The investigators will model the incremental costs and cost-effectiveness of intervention relative to standard-of-care TB diagnostic evaluation from the health system and patient perspective. The investigators will then construct an epidemic model of the population-level impact of the intervention strategy on TB incidence and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Site-level: Use standard (multi-day) sputum smear microscopy as the primary method of TB diagnosis
* Site-level: Participate in NTP-sponsored external quality assurance (EQA) for sputum smear microscopy
* Site-level: Send samples to a district or regional hospital/health center for Xpert testing
* Patient-level: Initiate evaluation for active TB at a study health center

Exclusion Criteria:

* Site-level: Do not agree to be randomized to standard-of-care vs. intervention arms
* Site-level: Perform sputum smear examination on <150 patients per year (based on 2015 data)
* Site-level: Diagnose <15 smear-positive TB cases per year (based on 2015 data)
* Patient-level: Have sputum collected for monitoring of response to anti-TB therapy
* Patient-level: Have sputum collected as part of active, community-based case finding (e.g., contact tracing, community outreach campaign)
* Patient-level: Referred to a study health center for TB treatment after a diagnosis is established elsewhere
* Patient-level: Started on TB treatment for extra-pulmonary TB only

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10644 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2022-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adithya Cattamanchi, MD, Principal Investigator — University of California, San Francisco
Locations (20):
- Uganda (20):
  - St Francis Njeru Health Center III, Buikwe
  - Busana Health Center III, Busana
  - Busesa Health Center IV, Busesa
  - Buwama Health Center III, Buwama
  - Iganga TC, Iganga
  - Bukulula Health Center IV, Kalungu
  - Nazigo Health Center III, Kayunga
  - Kiganda Health Center IV, Kiganda
  - Kira Health Center III, Kira
  - Lugasa Health Center III, Lugala
  - Bishop Asili Health Center, Luwero
  - Kinoni Health Center III, Lwengo
  - Kityerera Health Center IV, Mayuge
  - Malongo Health Center III, Mayuge
  - Mayuge Health Center III, Mayuge
  - Wabulungu Health Center III, Mayuge
  - Malangala Health Center III, Mityana
  - Lwampanga Health Center III, Nakasongola
  - Namungalwe Health Center III, Namungalwe
  - Nankandulo Health Center IV, Nankandulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] MacPherson P, Houben RM, Glynn JR, Corbett EL, Kranzer K. Pre-treatment loss to follow-up in tuberculosis patients in low- and lower-middle-income countries and high-burden countries: a systematic review and meta-analysis. Bull World Health Organ. 2014 Feb 1;92(2):126-38. doi: 10.2471/BLT.13.124800. Epub 2013 Nov 22. PMID 24623906
- [Background] Cattamanchi A, Dowdy DW, Davis JL, Worodria W, Yoo S, Joloba M, Matovu J, Hopewell PC, Huang L. Sensitivity of direct versus concentrated sputum smear microscopy in HIV-infected patients suspected of having pulmonary tuberculosis. BMC Infect Dis. 2009 May 6;9:53. doi: 10.1186/1471-2334-9-53. PMID 19419537
- [Background] Chihota VN, Ginindza S, McCarthy K, Grant AD, Churchyard G, Fielding K. Missed Opportunities for TB Investigation in Primary Care Clinics in South Africa: Experience from the XTEND Trial. PLoS One. 2015 Sep 18;10(9):e0138149. doi: 10.1371/journal.pone.0138149. eCollection 2015. PMID 26383102
- [Background] Davis J, Katamba A, Vasquez J, Crawford E, Sserwanga A, Kakeeto S, Kizito F, Dorsey G, den Boon S, Vittinghoff E, Huang L, Adatu F, Kamya MR, Hopewell PC, Cattamanchi A. Evaluating tuberculosis case detection via real-time monitoring of tuberculosis diagnostic services. Am J Respir Crit Care Med. 2011 Aug 1;184(3):362-7. doi: 10.1164/rccm.201012-1984OC. Epub 2011 Mar 11. PMID 21471088
- [Background] Aspler A, Menzies D, Oxlade O, Banda J, Mwenge L, Godfrey-Faussett P, Ayles H. Cost of tuberculosis diagnosis and treatment from the patient perspective in Lusaka, Zambia. Int J Tuberc Lung Dis. 2008 Aug;12(8):928-35. PMID 18647453
- [Background] Kemp JR, Mann G, Simwaka BN, Salaniponi FM, Squire SB. Can Malawi's poor afford free tuberculosis services? Patient and household costs associated with a tuberculosis diagnosis in Lilongwe. Bull World Health Organ. 2007 Aug;85(8):580-5. doi: 10.2471/blt.06.033167. PMID 17768515
- [Background] Simwaka BN, Bello G, Banda H, Chimzizi R, Squire BS, Theobald SJ. The Malawi National Tuberculosis Programme: an equity analysis. Int J Equity Health. 2007 Dec 31;6:24. doi: 10.1186/1475-9276-6-24. PMID 18163918
- [Background] Botha E, den Boon S, Lawrence KA, Reuter H, Verver S, Lombard CJ, Dye C, Enarson DA, Beyers N. From suspect to patient: tuberculosis diagnosis and treatment initiation in health facilities in South Africa. Int J Tuberc Lung Dis. 2008 Aug;12(8):936-41. PMID 18647454
- [Background] Ouyang H, Chepote F, Gilman RH, Moore DA. Failure to complete the TB diagnostic algorithm in urban Peru: a study of contributing factors. Trop Doct. 2005 Apr;35(2):120-1. doi: 10.1258/0049475054037002. No abstract available. PMID 15970047
- [Background] Steingart KR, Schiller I, Horne DJ, Pai M, Boehme CC, Dendukuri N. Xpert(R) MTB/RIF assay for pulmonary tuberculosis and rifampicin resistance in adults. Cochrane Database Syst Rev. 2014 Jan 21;2014(1):CD009593. doi: 10.1002/14651858.CD009593.pub3. PMID 24448973
- [Background] Dowdy DW, Cattamanchi A, Steingart KR, Pai M. Is scale-up worth it? Challenges in economic analysis of diagnostic tests for tuberculosis. PLoS Med. 2011 Jul;8(7):e1001063. doi: 10.1371/journal.pmed.1001063. Epub 2011 Jul 26. PMID 21814496
- [Background] Keeler E, Perkins MD, Small P, Hanson C, Reed S, Cunningham J, Aledort JE, Hillborne L, Rafael ME, Girosi F, Dye C. Reducing the global burden of tuberculosis: the contribution of improved diagnostics. Nature. 2006 Nov 23;444 Suppl 1:49-57. doi: 10.1038/nature05446. No abstract available. PMID 17159894
- [Background] Theron G, Zijenah L, Chanda D, Clowes P, Rachow A, Lesosky M, Bara W, Mungofa S, Pai M, Hoelscher M, Dowdy D, Pym A, Mwaba P, Mason P, Peter J, Dheda K; TB-NEAT team. Feasibility, accuracy, and clinical effect of point-of-care Xpert MTB/RIF testing for tuberculosis in primary-care settings in Africa: a multicentre, randomised, controlled trial. Lancet. 2014 Feb 1;383(9915):424-35. doi: 10.1016/S0140-6736(13)62073-5. Epub 2013 Oct 28. PMID 24176144
- [Background] Glasgow RE, Vogt TM, Boles SM. Evaluating the public health impact of health promotion interventions: the RE-AIM framework. Am J Public Health. 1999 Sep;89(9):1322-7. doi: 10.2105/ajph.89.9.1322. PMID 10474547
- [Background] Godin G, Belanger-Gravel A, Eccles M, Grimshaw J. Healthcare professionals' intentions and behaviours: a systematic review of studies based on social cognitive theories. Implement Sci. 2008 Jul 16;3:36. doi: 10.1186/1748-5908-3-36. PMID 18631386
- [Background] Davis DA, Thomson MA, Oxman AD, Haynes RB. Evidence for the effectiveness of CME. A review of 50 randomized controlled trials. JAMA. 1992 Sep 2;268(9):1111-7. PMID 1501333
- [Background] Cattamanchi A, Miller CR, Tapley A, Haguma P, Ochom E, Ackerman S, Davis JL, Katamba A, Handley MA. Health worker perspectives on barriers to delivery of routine tuberculosis diagnostic evaluation services in Uganda: a qualitative study to guide clinic-based interventions. BMC Health Serv Res. 2015 Jan 22;15:10. doi: 10.1186/s12913-014-0668-0. PMID 25609495
- [Background] Ivers N, Jamtvedt G, Flottorp S, Young JM, Odgaard-Jensen J, French SD, O'Brien MA, Johansen M, Grimshaw J, Oxman AD. Audit and feedback: effects on professional practice and healthcare outcomes. Cochrane Database Syst Rev. 2012 Jun 13;2012(6):CD000259. doi: 10.1002/14651858.CD000259.pub3. PMID 22696318
- [Background] Grogan S, Conner M, Norman P, Willits D, Porter I. Validation of a questionnaire measuring patient satisfaction with general practitioner services. Qual Health Care. 2000 Dec;9(4):210-5. doi: 10.1136/qhc.9.4.210. PMID 11101705
- [Background] Nabbuye-Sekandi J, Makumbi FE, Kasangaki A, Kizza IB, Tugumisirize J, Nshimye E, Mbabali S, Peters DH. Patient satisfaction with services in outpatient clinics at Mulago hospital, Uganda. Int J Qual Health Care. 2011 Oct;23(5):516-23. doi: 10.1093/intqhc/mzr040. Epub 2011 Jul 19. PMID 21775313
- [Background] Ivers NM, Halperin IJ, Barnsley J, Grimshaw JM, Shah BR, Tu K, Upshur R, Zwarenstein M. Allocation techniques for balance at baseline in cluster randomized trials: a methodological review. Trials. 2012 Aug 1;13:120. doi: 10.1186/1745-6215-13-120. PMID 22853820
- [Background] Sismanidis C, Moulton LH, Ayles H, Fielding K, Schaap A, Beyers N, Bond G, Godfrey-Faussett P, Hayes R. Restricted randomization of ZAMSTAR: a 2 x 2 factorial cluster randomized trial. Clin Trials. 2008;5(4):316-27. doi: 10.1177/1740774508094747. PMID 18697846
- [Background] Sandelowski M, Leeman J. Writing usable qualitative health research findings. Qual Health Res. 2012 Oct;22(10):1404-13. doi: 10.1177/1049732312450368. Epub 2012 Jun 28. PMID 22745362
- [Background] Sandelowski MJ. Justifying qualitative research. Res Nurs Health. 2008 Jun;31(3):193-5. doi: 10.1002/nur.20272. No abstract available. PMID 18288640
- [Background] Voils CI, Sandelowski M, Barroso J, Hasselblad V. Making Sense of Qualitative and Quantitative Findings in Mixed Research Synthesis Studies. Field methods. 2008;20(1):3-25. doi: 10.1177/1525822X07307463. PMID 18677415
- [Background] Salje H, Andrews JR, Deo S, Satyanarayana S, Sun AY, Pai M, Dowdy DW. The importance of implementation strategy in scaling up Xpert MTB/RIF for diagnosis of tuberculosis in the Indian health-care system: a transmission model. PLoS Med. 2014 Jul 15;11(7):e1001674. doi: 10.1371/journal.pmed.1001674. eCollection 2014 Jul. PMID 25025235
- [Background] Dowdy DW, Basu S, Andrews JR. Is passive diagnosis enough? The impact of subclinical disease on diagnostic strategies for tuberculosis. Am J Respir Crit Care Med. 2013 Mar 1;187(5):543-51. doi: 10.1164/rccm.201207-1217OC. Epub 2012 Dec 21. PMID 23262515
- [Background] Sun AY, Denkinger CM, Dowdy DW. The impact of novel tests for tuberculosis depends on the diagnostic cascade. Eur Respir J. 2014 Nov;44(5):1366-9. doi: 10.1183/09031936.00111014. Epub 2014 Sep 3. PMID 25186263
- [Background] Chandrasekaran V, Ramachandran R, Cunningham J, Balasubramaniun R, Thomas A, Sudha G, et al. Factors leading to tuberculosis diagnostic drop-out and delayed treatment initiation in Chennai, India. Int J Tuberc Lung Dis. 2005;9:172.
- [Background] Den Boon S, Semitala F, Cattamanchi A, Walter N, Worodria W, Joloba M, Huang L, Davis JL. Impact of patient drop-out on the effective sensitivity of smear microscopy strategies. Am J Respir Crit Care Med 2010;181:A2258.
- [Background] Miller C, Haguma P, Ochom E, Ross J, Davis JL, Cattamanchi A, Katamba A. Costs associated with tuberculosis evaluation in rural Uganda. 43rd Union World Conference on Lung Health; Kuala Lumpur, Malaysia 2012.
- [Background] WHO. Global strategy and targets for tuberculosis prevention, care and control after 2015. Geneva, Switzerland: World Health Organization, 2013 EB134/12.
- [Background] WHO. WHO monitoring of Xpert MTB/RIF roll-out. Available at: http://www.who.int/tb/areas-of-work/laboratory/mtb-rif-rollout/en/ [cited 2015 January 15].
- [Background] Churchyard GJ, on behalf of the Xtend study team. Xpert MTB/RIF vs microscopy as the first line TB test in South Africa: mortality, yield, initial loss to follow up and proportion treated. The Xtend Study. Conference on Retroviruses and Opportunistic Infections; Boston, USA: Available at: http://www.stoptb.org/wg/gli/assets/documents/M6/Churchyard%20-%20XTEND%20study.pdf; 2014.
- [Background] Cepheid. GeneXpert Omni: The True Point of Care Molecular Diagnostic System: Cepheid Inc; 2015. Available from: http://www.cepheid.com/us/genexpert-omni.
- [Background] Ajzen I. The theory of planned behavior. Organizational Behavior and Human Decision Processes. 1991;50:179-211.
- [Background] Green LW, Krueter M. Health Program Planning - An Educational and Ecological Approach. 4th ed. Philadelphia, USA: McGraw-Hill; 2005.
- [Background] Hayes RJ, Moulton LH. Cluster Randomized Trials. Boca Raton, Florida, USA: CRC Press; 2009.
- [Derived] Cattamanchi A, Reza TF, Nalugwa T, Adams K, Nantale M, Oyuku D, Nabwire S, Babirye D, Turyahabwe S, Tucker A, Sohn H, Ferguson O, Thompson R, Shete PB, Handley MA, Ackerman S, Joloba M, Moore DAJ, Davis JL, Dowdy DW, Fielding K, Katamba A. Multicomponent Strategy with Decentralized Molecular Testing for Tuberculosis. N Engl J Med. 2021 Dec 23;385(26):2441-2450. doi: 10.1056/NEJMoa2105470. PMID 34936740
- [Derived] Reza TF, Nalugwa T, Farr K, Nantale M, Oyuku D, Nakaweesa A, Musinguzi J, Vangala M, Shete PB, Tucker A, Ferguson O, Fielding K, Sohn H, Dowdy D, Moore DAJ, Davis JL, Ackerman SL, Handley MA, Katamba A, Cattamanchi A. Study protocol: a cluster randomized trial to evaluate the effectiveness and implementation of onsite GeneXpert testing at community health centers in Uganda (XPEL-TB). Implement Sci. 2020 Apr 21;15(1):24. doi: 10.1186/s13012-020-00988-y. PMID 32316993

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Community Health Centers
Groups:
- Intervention: Onsite molecular testing for TB with GeneXpert + process redesign to facilitate same-day TB diagnosis and treatment + performance feedback
  GeneXpert: Onsite molecular testing with GeneXpert as a replacement for microscopy
  Process re-design: Research and Uganda NTLP staff will engage health center staff in a discussion of how to re-organize clinical, laboratory and pharmacy services to enable same-day TB diagnosis and treatment.
  Performance Feedback: Feedback of TB diagnostic evaluation quality indicators to health center staff
Period: Overall Study
Arm/Group | Control Group | Intervention
Started | 5098; 10 Community Health Centers | 5546; 10 Community Health Centers
Completed | 5098; 10 Community Health Centers | 5546; 10 Community Health Centers
Not Completed | 0; 0 Community Health Centers | 0; 0 Community Health Centers

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Intervention | Total
Number analyzed (Participants) | 5098 | 5546 | 10644
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 38 [27 to 50] | 40 [30 to 52] | 40 [29 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3112 | 3289 | 6401
  Male | 1986 | 2257 | 4243
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5098 | 5546 | 10644
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5098 | 5546 | 10644
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 5098 | 5546 | 10644
HIV infection [Count of Participants; unit: Participants] — Population: Excludes participants with unknown HIV status
  Participants
    number analyzed (Participants) | 4290 | 5273 | 9563
    (all) | 1905 | 2285 | 4190

OUTCOME MEASURES:

1. Primary Outcome: Number Treated for Microbiologically-confirmed TB Within 14 Days After Presentation to the Health Center for TB Evaluation
Description: Effectiveness outcome.
Time Frame: Within 14 days after presentation to the health center for tuberculosis evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 5098 | 5546
Participants | 220 | 342
Statistical Analysis 1: Comparison: Control Group vs Intervention; Test type: Superiority; Rate Ratio (adjusted) = 1.56, 95% CI 2-sided [1.21 to 2.01]

2. Secondary Outcome: Number Diagnosed With Microbiologically-confirmed TB
Description: Effectiveness outcome.
Time Frame: Within 14 days after presentation to the health center for tuberculosis evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 5098 | 5546
Participants | 299 | 389
Statistical Analysis 1: Comparison: Control Group vs Intervention; Test type: Superiority; Rate Ratio (adjusted) = 1.28, 95% CI 2-sided [0.99 to 1.66]

3. Secondary Outcome: Time to Microbiologically-confirmed TB
Description: Effectiveness outcome. Time-to-diagnosis if microbiologically-confirmed TB.
Time Frame: Within 6 months of presentation to the health center for tuberculosis evaluation
Population: All participants' data was analyzed to determine who had confirmed TB.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 311 | 391
days | 0 [0 to 3] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Control Group vs Intervention; Test type: Superiority; Geometric Mean Ratio (adjusted) = 0.49, 95% CI 2-sided [0.39 to 0.62]

4. Secondary Outcome: Number Treated for TB
Description: Effectiveness outcome.
Time Frame: Within 14 days of presentation to the health center for tuberculosis evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 5098 | 5546
Participants | 339 | 485
Statistical Analysis 1: Comparison: Control Group vs Intervention; Test type: Superiority; Rate Ratio (adjusted) = 1.48, 95% CI 2-sided [1.04 to 2.12]

5. Secondary Outcome: Time-to-treatment of Microbiologically-confirmed TB
Description: Effectiveness outcome. Time-to-treatment if microbiologically-confirmed TB and treated.
Time Frame: Days from initial health center visit to initiation of treatment if diagnosed, up to 6 months.
Population: All participants' data was analyzed to determine who had confirmed TB and treatment initiated.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 267 | 351
days | 1 [0 to 8] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Control Group vs Intervention; Test type: Superiority; Geometric Mean Ratio (adjusted) = 0.35, 95% CI 2-sided [0.21 to 0.56]

6. Secondary Outcome: Number Who Died Within 6 Months
Description: Effectiveness outcome.
Time Frame: Within 6 months of presentation to the health center for tuberculosis evaluation
Population: Includes those with vital status follow-up at six months post-visit to health center
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 3695 | 4421
Participants | 123 | 116
Statistical Analysis 1: Comparison: Control Group vs Intervention; Test type: Superiority; Risk Ratio (RR) = 0.77, 95% CI 2-sided [0.44 to 1.35]

7. Secondary Outcome: Number of Patients Enrolled
Description: Effectiveness outcome.
Time Frame: Presentation to the health center for tuberculosis evaluation during the 16-month study time frame
Population: All eligible were enrolled as there was a waiver of informed consent
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 5098 | 5546
Participants | 5098 | 5546

8. Secondary Outcome: Number Tested for TB According to National Guidelines
Description: Effectiveness outcome.
Time Frame: Within 6 months of presentation to the health center for tuberculosis evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 5098 | 5546
Participants | 2687 | 5108

9. Secondary Outcome: Number Suspected/Diagnosed With Rifampin-resistant TB
Description: Effectiveness outcome.
Time Frame: Within 6 months of presentation to the health center for tuberculosis evaluation
Population: The data analyzed included all adult patients in the target population. Those with rifampin-resistant tuberculosis, extrapulmonary tuberculosis and/or missing age data were excluded from the trial population. Therefore, the number of participants analyzed for this measure differs from other parts of the record.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 5201 | 5637
Participants | 5 | 2

10. Secondary Outcome: Number Diagnosed and Treated for Microbiologically-confirmed TB
Description: Effectiveness outcome.
Time Frame: On the same-day of presentation to the health center for tuberculosis evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 5098 | 5546
Participants | 106 | 251

11. Secondary Outcome: Number Diagnosed AND Treated for TB
Description: Effectiveness outcome.
Time Frame: On the same-day of presentation to the health center for tuberculosis evaluation
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Intervention
Number analyzed (Participants) | 5098 | 5546
Participants | 199 | 362

ADVERSE EVENTS:
Time Frame: Vital status was assessed up to 18 months following health center visit
Description: For all-cause mortality, the denominator excludes those with unknown vital status and unknown HIV status. Vital status was ascertained through review of TB treatment registers, phone calls, and home visits.
  Serious and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Control Group | Intervention
All-Cause Mortality (participants affected / at risk) | 154/3857 | 145/4556
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT03044158/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/58/NCT03044158/ICF_001.pdf